CLINICAL TRIAL: NCT01720940
Title: Reducing Nephrotoxicity of Vancomycin: A Prospective, Randomized Study of Continuous Versus Intermittent Infusion of Vancomycin
Brief Title: Reducing Nephrotoxicity of Vancomycin: A Prospective Study of Continuous Versus Intermittent Infusion of Vancomycin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Medicine, Division of Infectious Diseases, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUHID-001
Record Dates: First submitted 2012-10-21; First posted 2012-11-02 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-11

CONDITIONS: Infections Requiring Prolonged Duration (>10 Days) of Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- continuous vancomycin infusion (Experimental)
  Interventions: Drug: continuous vancomycin infusion
- intermittent vancomycin infusion (Active Comparator): vancomycin in this arm will be administered as intermittent infusion
  Interventions: Drug: intermittent vancomycin infusion

INTERVENTIONS:
Drug: continuous vancomycin infusion — 24-hour continuous infusion of vancomycin
  Arms: continuous vancomycin infusion
Drug: intermittent vancomycin infusion
  Arms: intermittent vancomycin infusion

SUMMARY:
This study is being carried out to find out whether there is reduction in vancomycin-induced kidney injury (nephrotoxicity) when vancomycin is given as intermittent versus continuous infusion.

This study will recruit 220 subjects from 2 hospitals over a period of 3 years.

Participants are invited if they have an infection that requires prolonged vancomycin therapy (> more than 10 days).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 21-80 years
* Documented infection requiring prolonged (> 10 days) of vancomycin therapy
* Creatinine clearance > 50 ml/min (using Cockroft-Gault equation)

Exclusion Criteria:

* Patient already received 7 days or more of vancomycin therapy
* Pregnancy
* Severe burns > 40% body surface area
* Spinal cord injuries
* Participation in another interventional trial in previous 30 days
* Inability to obtain informed consent

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
nephrotoxicity | occurring any time while on vancomycin treatment up to 14 days post treatment completion
  nephrotoxicity as defined by the acute kidney injury network (AKIN) criteria using only serum creatinine criteria

SECONDARY OUTCOMES:
biomarkers for detection of early nephrotoxicity | measured weekly from the date of randomization until 14 days post completion of vancomycin
  serum and urine NGAL and cystatin C

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore